CLINICAL TRIAL: NCT06782048
Title: Pyrvinium for Reversal of Precancerous Metaplasia and Dysplasia in the Stomach
Brief Title: Use of Pyrvinium to Reverse Stomach Precancerous Conditions
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National University Hospital, Singapore (Other)
Collaborators: National University of Singapore (Other); Vanderbilt University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2024-3680
Record Dates: First submitted 2024-12-09; First posted 2025-01-17 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2024-12

CONDITIONS: STOMACH NEOPLASM
Keywords: Gastric Cancer; Stomach Neoplasm; Intestinal Metaplasia; Pyrvinium
MeSH Terms: conditions — Stomach Neoplasms | interventions — pyrvinium; Endoscopy, Digestive System; Biopsy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pyrvinium (Experimental): Pyrvinium will be administered to participants.
  Interventions: Drug: Pyrvinium; Procedure: Blood biomarkers analyses; Procedure: Oesophagogastroduodenoscopy (OGD) and biopsy; Other: Gastric juice, saliva and stool collection and analyses
- Placebo (Placebo Comparator): Placebo will be administered to participants.
  Interventions: Drug: Placebo; Procedure: Blood biomarkers analyses; Procedure: Oesophagogastroduodenoscopy (OGD) and biopsy; Other: Gastric juice, saliva and stool collection and analyses

INTERVENTIONS:
Drug: Placebo — Participants will receive placebo by mouth once each day for a total of 14 days.
  Arms: Placebo
Drug: Pyrvinium — Participants will receive pyrvinium (2 mg/kg/day) by mouth once each day for a total of 14 days.
  Arms: Pyrvinium
Procedure: Blood biomarkers analyses — Up to 20ml of blood will be drawn from each participant at each study visit, with a total of 4 study visits for molecular analyses.
Procedure: Oesophagogastroduodenoscopy (OGD) and biopsy — Study participant will undergo OGD with collection of gastric mucosal biopsies at the baseline visit to ascertain IM status and for molecular analyses. Study participant will undergo follow-up gastroscopy with collection of gastric mucosal biopsies at day 7 of treatment, 6 weeks post-treatment and 1 year post-treatment to assess if endpoint is reached and for molecular analyses. Gastric juice samples will be collected during each OGD.
Other: Gastric juice, saliva and stool collection and analyses — Gastric juice will be taken, and gastric pH will be measured at each research endoscopy. Saliva and stool will also be obtained from participants at research endoscopy for microbiome studies at the following timepoints: baseline, 6 weeks post-treatment, and 1 year post-treatment.

SUMMARY:
This study is carried out to find out if a drug called pyrvinium is able to convert pre-cancerous tissue in the stomach back to healthy tissue, to lower the chances of stomach cancer. Pyrvinium is a drug that has been used for a long time to treat pinworms in children and its anti-cancer properties are currently under investigation. Tests in animals have shown that pyrvinium made unhealthy tissue healthier and stopped some cells from growing in a bad way. Based on preclinical studies, the investigators hypothesise that the proportion of samples with pre-cancerous tissue in the stomach would decrease by 50% after exposure to pyrvinium at the 6-week timepoint, with anticipated durability of the response at the one-year follow-up.

DETAILED DESCRIPTION:
Objectives:

The main objectives of the study are to gain additional data on the efficacy and safety for the use of pyrvinium in human participants with gastric intestinal metaplasia and/or dysplasia for reversion to complete intestinal metaplasia or normal gastric mucosa. The secondary objectives are to evaluate effectiveness of pyrvinium treatment in human pre-cancerous gastroids derived from patients with metaplasia and/or dysplasia, determine targeted effects of pyrvinium treatment in heterogeneous pre-cancerous cells, define functional mechanisms of pyrvinium action as an anti-cancer drug, determine effects of pyrvinium on the level of serum biomarkers associated with GC risk prediction and investigate the impact of pyrvinium on the gastric microbiome.

Study Design:

This is a phase 2 randomized clinical trial which aims to recruit 50 participants with extensive/marked intestinal metaplasia (IM) and/or dysplasia. After enrolment, a baseline oesophagogastroduodenoscopy (OGD) is performed using a modified Cambridge protocol to ensure adequate sampling. As most participants will be recruited prior to confirming their histology at baseline, some participants will be withdrawn from the study if they are detected to have no IM, no extensive/marked IM, or no dysplasia at baseline. 50 participants with evidence of extensive/marked gastric IM and/or dysplasia will receive pyrvinium (2mg/kg/day) or placebo orally in a 1:1 randomization ratio daily for a period of 14 days. Participants will be followed up at the clinic or via telephone for monitoring of symptoms at Day 14 of treatment. Participants will remain blinded, and study team will be split into blinded and unblinded teams. Only the unblinded team will have access to exposure (pyrvinium vs placebo) during the active phase of the trial. In total, there will be 3 follow-up study visits at the clinic after randomization, for up to a year after the last day of treatment.

Baseline:

Participants will undergo a baseline OGD and biopsy to ascertain IM and dysplasia status. Gastric mucosal biopsies will be collected as follows:

* 1 biopsy each from AL, AG, IA, BL, BG, PP and sent for histological examination
* 3 adjacent biopsies at BL, 1 biopsy at IA, 5 adjacent biopsies at AL, 1 biopsy at AG and 2 adjacent biopsies at PP, will be snap-frozen in liquid nitrogen

The locations are defined as follows:

* AL - lesser curvature of the antrum, within 2-3cm of the pylorus
* AG - greater curvature of the antrum, within 2-3cm of the pylorus
* IA - incisura angularis
* BL - lesser curvature of the corpus, 4cm proximal to the angulus
* BG - middle portion of the greater curvature of the corpus, 8cm from the cardia
* PP - prepylorus

Gastric juice will be taken if there is an opportunity to do so, and gastric pH will be measured. 4 biopsies of areas of known gastric IM will be used to generate gastric organoids. Participants with evidence of extensive/marked gastric IM and/or dysplasia will then be randomized to either the pyrvinium or placebo treatment arm. Clinical data including co-morbidities, medication use, H. pylori testing and treatment history, family history, tobacco and alcohol exposures, endoscopic data, and pathology/histology results will be collected at the time of enrolment.

The initial IM lesion area is located by targeting EGGIM II, which correlates well with extensive IM. The gastric mucosa is observed with HD-WLE followed by HD-NBI. The OGD procedure will be recorded for verification purposes. All mucosal lesions identified during OGD will be biopsied separately as a part of normal clinical practice and sent for histopathological assessment. Frozen biopsy samples will be stored at a high-quality tissue bank. Investigators will follow the above protocol. However, they may deviate from protocol if the interests of the patient require so.

Histological Assessment:

For histological evaluation, biopsies will be stained for H&E as well as PAS/Alcian blue. In addition, immunostaining will be performed for markers of normal gastric lineages, metaplasia (SPEM and IM) and dysplasia. Marker expression in biopsies will be evaluated with digital imaging and quantitation.

Food Frequency Questionnaire (FFQ):

Participants will be asked to complete an FFQ once at the baseline visit, within 4 weeks from the stool sample collection.

Follow-up:

Both pyrvinium and placebo groups will undergo the same follow-up procedures. Mucosal biopsies will be collected at each of the follow-up surveillance OGDs as follows:

* 1 biopsy each from AL, AG, IA, BL, BG, PP and sent for histological examination
* 2 adjacent biopsies at BL, 4 adjacent biopsies at AL and 2 adjacent biopsies at PP will be snap-frozen in liquid nitrogen

A maximum of 14 research biopsies will be taken at each of the follow-up endoscopies. The EGGIM score will be recorded. The gastric mucosa is observed with HD-WLE followed by HD-NBI. The OGD procedure will be recorded for verification purposes. All mucosal lesions identified during OGD will be biopsied separately as a part of normal clinical practice and sent for histopathological assessment. Frozen biopsy samples will be stored at a high-quality tissue bank. Investigators will follow the above protocol. However, they may deviate from protocol if the interests of the patient require so.

Follow-up surveillance OGDs will be done at Day 7 of treatment, 6 weeks post-treatment and 1 year post-treatment. A window period of ± 2 days for the surveillance OGD at Day 7 of treatment, and ± 2 weeks for the surveillance OGD at 6 weeks and 1-year post-treatment are acceptable.

Symptoms will be monitored via clinic or telephone follow-up on the last day of the treatment (Day 14). Known rare side-effects include skin rash, sun-sensitivity, diarrhoea, nausea/vomiting, stomach cramps and these and other symptoms will be monitored in all subjects.

Blood Collection, Processing and Analyses:

Up to 20ml of blood will be drawn from each participant at each of the following timepoints: baseline, day 7 of treatment, 6 weeks post-treatment and 1 year post-treatment. The serum, plasma and buffy coat will be extracted.

Gastric Juice, Saliva and Stool Collection:

Gastric juice will be taken, and gastric pH will be measured at each research endoscopy, i.e., baseline, day 7 of treatment, 6 weeks post-treatment and 1 year post-treatment. Saliva and stool will also be obtained from participants at research endoscopy for microbiome studies at the following timepoints: baseline, 6 weeks post-treatment, and 1 year post-treatment.

Human Pre-cancer Organoids:

The investigators will perform biological studies using human organoids derived from patients recruited for the phase 2 clinical trial, with the aim of determining targeted effects of pyrvinium treatment in heterogeneous pre-cancerous cells and define functional mechanisms of pyrvinium action as an anti-cancer drug.

Serum Biomarker Profiling:

Total RNA from serum is isolated and converted to cDNA, which is then quantified. Target miRNA expression levels after normalization of both technical and biological variations are analysed to identify panels of miRNAs with the highest discriminatory power between healthy and disease states.

Microbiota Analyses:

Tissues, gastric juice, saliva and stool will undergo next generation metagenomic sequencing and directed culturomics, to study microbe-host interactions in IM progression/regression.

Single Cell Analysis:

Tissues will be placed into cold tissue storage solution and dissociated into single cells using enzymatic digestion and trypan blue staining will be performed to determine cell viability. Dissociated cells will then be used for various single cell platforms such as scRNA-seq, scDNA-seq, scATAC-seq, single-cell immune profiling and other single-cell related technologies (accompanied by in- depth integrative computational data analysis) to determine the respective biological measurements. In addition to this, tissues might also be used for several genomic platforms (eg. exome sequencing and low pass sequencing etc) and immunohistological platforms.

Sample Size Calculation:

A sample size of 48 participants (24 per group) will be required to detect a difference of 30% in proportion of participants with a reduction in gastric intestinal metaplasia (primary endpoint) between the treatment (Pyrvinium) and control (Placebo) groups to achieve 80% power at 20% one-side type-I error rate, assuming close to 0% participants will have any reduction in gastric intestinal metaplasia, and 20% potential drop-out rate. The study design is referred to as Phase II Screening Trial Design, which has 80% chance to detect the treatment is truly effective and worth investigating further in a Phase III trial if the study results favourable to the treatment. The recruitment target has been rounded up from 48 to 50 participants.

Statistical Analysis:

(A) General considerations

The investigators hypothesise that pyrvinium (oral 2mg/kg/day for 14 days) compared to the control placebo would result in an absolute 50% reduction in gastric IM, whereby our advanced gastric IM patients have a mean 75.6% +/- 8.4%(SD) presence of IM in their biopsies compared to mild gastric IM patients with a mean 14% +/- 8.2%(SD) presence of IM in their gastric biopsies.

Continuous variables will be summarized using descriptive statistics including means, medians, Q1 and Q3, minimum and maximum, and standard deviations. Categorical variables will be summarized using percentages and frequencies. All confidence intervals are 95%.

(B) Efficacy analyses

All efficacy analysis will be performed based on the intention-to-treat population. The primary endpoint of percentage of patients with a reduction in gastric intestinal metaplasia (and/or dysplasia for reversion to complete intestinal metaplasia or normal gastric mucosa) will be calculated for the treatment and placebo group separately. The difference in the percentage will be presented along with 95% exact confidence interval. No p-values will be reported considering exploratory nature of the study. Secondary endpoints with binary outcomes will be analysed similar to the primary endpoint. Secondary continuous endpoints will be presented as mean change from baseline at the follow-up time-points. The difference in mean values between the groups will be presented at each follow-up time-point along with their 95% confidence intervals.

(C) Safety analyses

All safety analysis will be presented based on the treated population. Adverse and serious adverse events will be presented with number of subjects experiencing each type of adverse events and serious adverse events along with their relationship with the group and severity using counts and percentages. Laboratory results will be presented with their mean values at each assessment time-points along with the percentage of abnormal and clinically significant results for each group.

(D) Interim analyses

There is no formal interim analysis planned. However, the Principal Investigator will monitor the safety data in a blinded manner periodically. There would be periodic monitoring of the safety data by a committee comprising the NUH Endoscopy Centre Director, NUH Gastroenterology and Hepatology Head of Department, and NUH Gastroenterology and Hepatology Department Safety Lead.

ELIGIBILITY:
Inclusion Criteria:

* The subject is at least 21 years of age.
* The subject has histologically proven extensive/marked intestinal metaplasia and/or dysplasia.
* The subject is willing and able to provide signed and dated patient informed consent form indicating that he/she has been informed of all pertinent aspects of the study.

Exclusion Criteria:

* The subject has an active gastric cancer diagnosis.
* The subject is pregnant.
* The subject has a high-risk of bleeding complications due to anticoagulants or underlying medical condition such as bleeding disorders in whom biopsies are contraindicated.
* The subject has impaired renal function.
* The subject has impaired hepatic function.
* The subject has fructose intolerance, glucose-galactose malabsorption or sucrase-isomaltase deficiency.
* The subject has chronic bowel disease.
* The subject has any other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may interfere with the interpretation of study results and in the judgement of the investigator would make the subject unsuitable for entry into the study.
* The subject is unwilling or unable to provide signed informed consent.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-08 (Estimated); Primary Completion 2029-12 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Histological Regression of GIM: Average percentage change of GIM in the antrum and corpus, as measured by histological evaluation of gastric biopsies at baseline and the study endpoint | Baseline, 6 weeks post-treatment

SECONDARY OUTCOMES:
Surface Area of GIM Involvement: Measured in real-time using AI-guided imaging technology during endoscopy | During endoscopy at baseline, Day 7 of treatment, 6 weeks post-treatment and 1 year post-treatment
Safety: Number of participants with treatment-related adverse events | From Day 1 to Day 14 of treatment
Efficacy in Patient-Derived Gastroids: Changes in phosphorylation levels of proteins in pre-cancerous gastroids derived from participants with GIM or dysplasia | Baseline
  A maximum of 18 research biopsies will be taken at the baseline endoscopy, of which 4 biopsies of areas of known gastric IM will be used to generate gastric organoids.
Efficacy in Patient-Derived Gastroids: Evaluation of growth and proliferation after pyrvinium treatment via imaging, staining and histological techniques | Baseline
  A maximum of 18 research biopsies will be taken at the baseline endoscopy, of which 4 biopsies of areas of known gastric IM will be used to generate gastric organoids.
Mechanistic Insights into Pyrvinium Action: Gene expression profiles (e.g., mucins MUC1, MUC2, MUC5AC) in biopsied gastric samples obtained during endoscopy | Baseline, Day 7, 6 weeks post-treatment, 1 year post-treatment
Serum Biomarkers for Gastric Cancer Risk: Levels of serum biomarkers such as TFF3, a known marker for gastric IM, measured via ELISA | Baseline, Day 7 of treatment, 6 weeks post-treatment, 1 year post-treatment
Impact on Gastric Microbiome: Changes in gastric microbiome composition post-treatment, analyzed using advanced sequencing methods | Baseline, 6 weeks post-treatment, 1 year post-treatment

CONTACTS AND LOCATIONS:
Locations (1):
- National University Hospital, Singapore, Singapore